CLINICAL TRIAL: NCT06611722
Title: A Clinical Retrospective Cross-sectional Study of the Differences in the Psychological States of Patients with Different Chronic Hip Pain
Brief Title: The Differences in the Psychological States of Patients with Different Chronic Hip Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: ChunBao Li (Other)
Responsible Party: Sponsor-Investigator, ChunBao Li, deputy chief physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: 2023KY031-KS001
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Psychological Disorders; Hip Pain Chronic
Keywords: hip; pain; Psychological Disorders; depression; anxiety
MeSH Terms: conditions — Mental Disorders; Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- intra-articular hip pain group
  Interventions: Other: Psychological and Functional Assessment
- extra-articular hip pain group
  Interventions: Other: Psychological and Functional Assessment
- intra-articular combined extra-articular hip pain group
  Interventions: Other: Psychological and Functional Assessment

INTERVENTIONS:
Other: Psychological and Functional Assessment — Assessment of Pain Sources: Patients are grouped based on intra-articular, extra-articular, or combined intra- and extra-articular hip pain.Psychological Assessment: Depression and anxiety are assessed using standardized questionnaires (e.g., BDI for depression, SAS for anxiety).Functional Assessment: Joint function and pain are evaluated using clinical and patient-reported outcome measures.

SUMMARY:
Nowadays, studies related to the psychological state of patients with chronic hip pain are still limited, and there is a lack of research on the characteristics of the psychological state of patients with chronic soreness from different pain sources. The goal of this retrospective cross-sectional study was to reveal differences between the psychological states of chronic hip pain patients with different pain sources. The main question it aims to answer is whether there are differences in psychological states among hip pain patients with intra-hip pain, extra-hip pain, and intra-hip combined with extra-hip pain.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 16 years old and of sound mind；
* Chronic hip pain persisting for a duration exceeding 3 months.

Exclusion Criteria:

* Previous mental illness and cognitive impairment；
* Other serious illnesses such as heart failure, respiratory failure, malignant tumours, severe trauma and other serious illnesses;；
* Chronic pain lasting for more than 3 months in other parts of the body;；
* Use of prescribed opioid drugs exceeding 60 mg morphine equivalent per day or steroid analgesics.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic hip pain who visited the hip joint specialist outpatient clinic of the PLA General Hospital were included in the study. The diagnosis was made by the same docter based on clinical and radiological examinations, with a clear diagnosis of hip disease. Patients were divided into three groups according to the source of pain: intra-articular pain group, extra-articular pain group, and intra-articular combined extra-articular pain group. Intra-articular hip pain encompasses a range of conditions, including femoral acetabular impingement (FAI) and labral damage within the hip joint. Extra-articular hip pain encompasses conditions such as trochanteric bursitis and gluteal fasciitis. Combined hip pain represents a combination of both of these etiological factors.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
the Beck Depression Inventory (BDI) | 5 minutes
  The BDI is a self-assessment scale that has been demonstrated to be a reliable and valid tool for evaluating depressive symptoms. The BDI comprises 21 items, each item is assigned a score on a scale of 0 to 3, with higher scores indicating a greater severity of depressive symptoms.
the Zung Self-Rating Anxiety Scale (SAS) | 5 minutes
  The SAS is a self-assessment instrument designed to evaluate the presence and severity of anxiety symptoms. The SAS consists of 20 items, each item consisting of four statements, and each item is scored on a scale of 1 to 4. A higher score indicates a higher level of anxiety.

SECONDARY OUTCOMES:
the Visual Analogue Scale (VAS) | 2 minutes
  for the assessment of the level of hip pain perceived by the patient
the Pain Sensitivity Questionnaire (PSQ) | 5 minutes
  for the assessment of the individual's sensitivity to pain
The Hip Outcome Score Activities of Daily Living (HOS-ADL) | 5 minutes
  evaluate the functional activities necessitated by daily life with the hip
The Hip Outcome Score - Sport-specific subscale (HOS-SSS) | 5 minutes
  assess the capacity to perform sports activities
the modified Harris Hip Score (mHHS) | 5 minutes
  assess the functional level of the hip joint
the international hip outcome tool (IHOT-12) | 5 minutes
  assess the functional level of the hip joint

CONTACTS AND LOCATIONS:
Overall Officials: Chunbao Li, Study Director — The Fourth Medical Centre of the General Hospital of the People's Liberation Army
Locations (1):
- General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality, China